CLINICAL TRIAL: NCT04389281
Title: Phase 1 Study of X-PACT (X-ray Psoralen Activated Cancer Therapy) for Intra-tumoral Injection of Superficial Tumors in Patients With Advanced Head and Neck Cancer, Breast Cancer, Soft Tissue Sarcoma or Melanoma
Brief Title: X-ray Psoralen Activated Cancer Therapy in Head and Neck, Breast, Sarcoma and Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immunolight, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X-PACT 101
Record Dates: First submitted 2020-05-04; First posted 2020-05-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor Cancer
Keywords: Advanced Head & Neck Cancer; Advanced Breast Cancer; Advanced Melanoma; Advanced Soft Tissue Sarcoma; Advanced Solid Tumor
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Part One - Single Group, Open Label - Solid Tumor
  Part Two - Randomized to either 10 or 14 X-PACT treatments with either 1.35 or 2.0 Gy of radiation and to active the study drug and single or double phosphor administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Solid Tumor Cohort (Experimental): Single Arm (Part I): Open Label Solid Tumor Study: single arm consisting of a six-week treatment period with X-PACT (phosphor device and methoxsalen sterile solution and subsequently exposing the tumor to X-ray energy) administered as an intra-tumoral injection. Up to 7 X-PACT treatments will be administered at 1x phosphors and 1.35 Gy Radiation
  Interventions: Combination Product: X-PACT
- Expansion Cohort - 10 Treatments, 1x Phosphors, 2 Gy Radiation (Active Comparator): Randomized (Part II) - 4 patient Soft Tissue Sarcoma cohort and a 4 patient Triple Negative Breast Cancer cohort.
  Arm 1 - 10 X-PACT Treatments, 1x phosphors/tumor volume, 2.0 Gy Radiation
  Interventions: Combination Product: X-PACT
- Expansion Cohort - 14 Treatments, 1x Phosphors, 2 Gy Radiation (Active Comparator): Randomized (Part II) - 4 patient Soft Tissue Sarcoma cohort and a 4 patient Triple Negative Breast Cancer cohort.
  Arm 2 - 14 X-PACT Treatments, 1x phosphors/tumor volume, 2.0 Gy Radiation
  Interventions: Combination Product: X-PACT
- Expansion Cohort - 10 Treatments, 2x Phosphors, 1.35 Gy Radiation (Active Comparator): Randomized (Part II) - 4 patient Soft Tissue Sarcoma cohort and a 4 patient Triple Negative Breast Cancer cohort.
  Arm 3 - 10 X-PACT Treatments, 2x phosphors/tumor volume, 1.35 Gy Radiation
  Interventions: Combination Product: X-PACT
- Expansion Cohort - 14 Treatments, 2x Phosphors, 1.35 Gy Radiation (Active Comparator): Randomized (Part II) - 4 patient Soft Tissue Sarcoma cohort and a 4 patient Triple Negative Breast Cancer cohort.
  Arm 4 - 14 X-PACT Treatments, 2x phosphors/tumor volume, 1.35 Gy Radiation
  Interventions: Combination Product: X-PACT

INTERVENTIONS:
Combination Product: X-PACT — X-PACT is comprised of a phosphor device, the drug methoxsalen sterile solution and X-ray energy. The dose of methoxsalen sterile solution per injection will vary per patient and will remained fixed across injections within each patient as it is based on the applicable tumor volume at baseline. Immediately after each injection of the combination product, patients will be exposed to an X-ray beam delivered via a LINAC (and thus targeted at the tumor) at a fixed dose to activate the combination product.

SUMMARY:
In this Phase I trial for subjects with advanced head & neck cancer, breast cancer, soft tissue sarcoma or melanoma all subjects will receive open label X-PACT treatment as a intra-tumoral injection. The primary objective will be to establish the safety of X-PACT when dosed with 5 intra-tumoral injections of the combination product (the phosphor device and methoxsalen sterile solution and subsequently exposing the tumor to X-ray energy) over a period of 6 weeks (on day D1, D3 and D5 of Week 1, on D1 of Week 2, and a booster on D1 of Week 6). After the week 8 tumor assessment subjects demonstrating stable disease, partial response or unconfirmed progression assessed by iRecist, will be eligible to receive two additional booster treatments 4-6 weeks apart. Treatment will be considered safe provided ≤ 2 out of 12 patients experience a dose-limiting toxicity (DLT) during the 6 weeks after the first intra-tumoral injection.

Two expansion cohorts have been added to the study. One for TNBC and one for soft tissue sarcoma. 16 additional subjects will be added in each of the expansion cohorts.

DETAILED DESCRIPTION:
The primary endpoint will be to establish the safety of X-PACT when dosed with 5 intra-tumoral injections of the combination product (the phosphor device and methoxsalen sterile solution and subsequently exposing the tumor to X-ray energy) over a period of 6 weeks (on day D1, D3 and D5 of Week 1, on D1 of Week 2, and a booster on D1 of Week 6). After the week 8 tumor assessment subjects demonstrating stable disease, partial response or unconfirmed progression assessed by iRecist, will be eligible to receive two additional booster treatments 4-6 weeks apart. Part C has been added to the study to allow patients who respond to treatment to receive an additional 12 treatments over 12 months. In part C, up to two tumors in up to two radiation fields may be treated. Treatment will be considered safe provided ≤ 2 out of 12 patients experience a dose-limiting toxicity (DLT) during the 6 weeks after the first intra-tumoral injection. Subjects will have staging scans at baseline, day 8, week 7 and as per standard of care during the optional treatment and follow up study periods. Patients will be followed until they are lost to follow-up, refuse further follow-up or until death.

Subjects in each of the expansion cohorts will be randomized to receive either 10 or 14 X-PACT treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent
3. ECOG Performance Status of ≤ 1
4. Subjects with histologically or cytologically confirmed advanced solid tumors which have progressed after standard therapy(ies), intolerant to standard therapy, refused standard therapy or for which no standard therapy(ies) exist. Furthermore, the tumor targeted for injections should be:

   1. A non-visceral tumor, a metastatic lymph node, a metastasis from a visceral solid tumor provided the lesion is extravisceral, or a cutaneous tumor. Visceral tumors will not be treated.
   2. The tumor must be measurable as per RECIST criteria.
   3. The tumor should be directly accessible for injection or accessible with the use of ultrasound/CT guidance.
   4. The tumor identified for injection should be selected so local control could potentially provide benefit to the patient.
   5. 80% of the tumor must be accessible for injection with X-PACT (assessed by the treating physician)
   6. The tumor must be superficial and not exceed a depth of 5 cm.
   7. Eye or brain tumors will not be treated.
5. A patient with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to day 1 of treatment, have been off of corticosteroids for ≥ 2 weeks, and brain metastases are asymptomatic.
6. The study site Radiation Oncologist Investigator/sub-investigator has determined additiional radiation delivered via X-PACT is appropriate given patient's prior radiation exposure. The treating Radiation Oncologist will review all prior radiation received to the proposed site of X-PACT treatment and assess the potential for unacceptable toxicity to the site or local organ(s) using QUANTEC.
7. All toxicities from prior therapy should be ≤Grade 1 before start of study treatment. All radiation associated toxicities must have completely resolved to be considered for inclusion into the study.
8. Demonstrate adequate organ function as defined in the table below:

   Hematological:

   White blood cell (WBC) ≥ 3 x 109/L Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L Platelet Count ≥ 100 x 109/L Hemoglobin (Hgb) ≥ 8 g/dL2

   Renal:

   Serum creatinine OR Creatinine clearance ≤ 1.5 x upper limit of normal (ULN) OR, in patients with a serum creatinine 1.5 x ULN, ≥ 60 mL/min as measured by a 24-hour urine collection or estimated by the Cockcroft and Gault formula

   Hepatic:

   Total bilirubin ≤ 1.5 × ULN (in patients with known Gilbert Syndrome a total bilirubin ≤3.0× ULN with direct bilirubin ≤1.5 X ULN) Aspartate aminotransferase (AST) ≤ 2.5 × ULN (or ≤ 5 if liver metastases are present) Alanine aminotransferase (ALT) ≤ 2.5 × ULN (or ≤ 5 if liver metastases are present)

   Coagulation:

   International Normalized Ratio (INR) ≤ 1.5
9. Females of childbearing potential (FCBP) must have a negative serum pregnancy test within 3 days prior to day 1 of treatment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
10. FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 28 days after treatment discontinuation. Contraceptive methods with low user dependency are preferable but not required (see table below, adapted from:

http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf)

Highly Effective Birth Control Methods:

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

  o oral
  * intravaginal
  * transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation

  o oral
  * injectable
  * implantable
* intrauterine device (IUD)
* intrauterine hormone-releasing system (IUS)
* vasectomised partner
* sexual abstinence

  11. Male patients must be willing to use condoms from the time of informed consent until 28 days after treatment discontinuation. For a non-pregnant FCBP partner, contraception recommendations should also be considered.

  12. As determined by the enrolling physician, ability of the patient to understand and comply with study procedures for the entire length of the study

  13. Patient is expected to have a life expectancy of at least 4 months

  14. If the proposed site of treatment with X-PACT had prior exposure to curative-intent radiation, the patient may be entered into the trial with the following provisions satisfied.
* There is at least a 6 month wash out period from the last date radiation was received to assess for radiation toxicity.
* If there was previous radiation toxicity at the proposed site of X-PACT, the toxicity resolved at least three months ago and the site did not involve a major organ.
* The site investigator in addition to the radiation oncologist (as a part of criterion #6) has fully reviewed the subject's radiation history, has examined the area for radiation toxicity and assessed the cumulative dose for either 5 or 7 X-PACT treatments and determined they will not pose additional risk for radiation toxicity or re-activate any other previous toxicity.

Exclusion Criteria:

* Exclusion Criteria:

  1. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study.)
  2. Prior exposure to methoxsalen
  3. History of any of the following:

     a. Idiosyncratic or hypersensitivity reactions to any psoralen compounds or any of their excipients

     b. Light sensitive disease state

     c. Disease associated with photosensitivity including lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum and albinism

     d. Aphakia
  4. History of idiosyncratic or hypersensitivity reactions to any of the phosphor device components
  5. Known diagnosis of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection (NOTE: testing not required)
  6. Active infection requiring systemic therapy (NOTE: at discretion of investigator, patients with uncomplicated urinary tract infections may be eligible.)
  7. Has a known additional other primary malignancy that is active and/or progressive requiring treatment; exceptions include basal cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the patient has been disease-free for at least five years.
  8. Systemic anti-cancer treatment within 28 days (or 5 half-lives, whichever is shorter) prior to day 1 of treatment
  9. Treatment with any investigational drug within 5 half-lives or 28 days, whichever is shorter (or if half-life is unknown, within 28 days) prior to day 1 of treatment
  10. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

      a. Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded)

      b. Uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 105 mmHg at screening) despite two concomitant antihypertensive therapies.

      c. Acute myocardial infarction or unstable angina ≤ 6 months prior to day 1 of treatment

      d. New York Heart Association Class III or IV congestive heart failure (
  11. Other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator.
  12. The tumor identified for treatment has a volume greater than 500 cc (Soft Tissue Sarcoma only). All other tumor types may have a maximum volume of 300 cc
  13. Receiving or planned use of corticosteroids. Subjects will require a one-week washout period from prior corticosteroid use. Inhaled or topical steroids are permitted.
  14. Subjects with active autoimmune disease requiring 10 mg or greater of prednisone and/or biologic agents.
  15. Subjects with a history of pancreatitis or elevated baseline serum lipase without otherwise specified etiology.

For the Expansion Cohorts, the inclusion criteria remain the same except for Inclusion Criteria #4 and #14 and which reads:

4. Subjects with histologically and/or cytologically confirmed, inoperable locally advanced, recurrent or metastatic triple-negative breast cancer* (TNBC Cohort) or advanced, metastatic or relapsed soft tissue sarcoma** (STS Cohort). Furthermore, the tumor targeted for injections should be:

1. A non-visceral tumor, a metastatic lymph node, a metastasis from a visceral solid tumor provided the lesion is extravisceral, or a cutaneous tumor. Visceral tumors will not be treated.
2. The tumor must be measurable as per RECIST criteria, at least 1 cm for masses and 1.5 cm for lymph nodes.
3. The tumor should be directly accessible for injection or accessible with the use of ultrasound/CT guidance.
4. 80% of the tumor must be accessible for injection with X-PACT (assessed by the treating physician)
5. Up to 4 target lesions may be selected for injection in up to two radiation fields, but the radiation fields may not overlap, however, the total phosphors delivered may not exceed 840 mg for each treatment day (e.g. investigators may elect to treat only one very large tumor, two medium tumors, one large and one small tumor, or 4 very small tumors to ensure the total phosphors limit per treatment). Selected lesions must represent at least 50% of the tumor load by investigator determination.

   * For the TNBC Cohort, participants must have either unresectable, locally advanced, relapsed, refractory or metastatic disease with HER2 negative/low ER/PR status (<10%) or HER2 negative/ER/PR negative. Patients determined to be HER2 ultra-low will not be enrolled. Furthermore, participants must have received at least one prior treatment (best medical treatment for cancer stage, PDL-1 status, BRCA 1 or 2 status and general health status) as per Figure 26-1 (see Protocol for schematic . Participants who are intolerant or refuse best medical care would also be eligible.

     * For the STS Cohort, participants must have received at least one prior treatment (best medical treatment recommended for the participants sub-type) for unresectable, locally advanced, relapsed, refractory or metastatic disease. Participants who are intolerant to or have refused best medical treatment for their subtype will also be eligible. Best medical treatment includes: surgery, radiation, chemotherapy (including doxorubicin, Trabectedin), gene therapy, targeted therapy (pazopanib) or antibody-drug conjugates.

       * 14 It is preferable to select tumors that have not been previously radiated, but if other options are not available and the tumor selected is in a field which received curative-intent radiation, then the participant may only be enrolled with the following provisions satisfied.

         * There is at least a 6 month wash out period from the last date radiation was received to assess for radiation toxicity.
         * If there was previous radiation toxicity at the proposed site of X-PACT, the toxicity resolved at least three months ago and the site did not involve a major organ.
         * The site investigator in addition to the radiation oncologist (as a part of criterion #6) has fully reviewed the subject's radiation history, has examined the area for radiation toxicity, has assessed the cumulative dose for total X-PACT treatments and determined they will not pose additional risk for radiation toxicity or re-activate any other previous toxicity.

For the TNBC cohort the following exclusion criteria has been added:

17. For the TNBC Cohort, patients determined to be HER2 ultra-low.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | First 6 weeks
  The primary objective will be to establish the safety of X-PACT when dosed at the schedule described above, with X-PACT considered safe provided ≤ 2 out of 12 patients experience a dose-limiting toxicity (DLT) during the 6 weeks after the first intra-tumoral injection.

SECONDARY OUTCOMES:
Evaluate Local Response Rate (LRR) | After first 6 weeks of treatment
  Evaluate local response rate by assessing treated tumor volume pre and post treatment
Evaluate Durability of Response | Post first 6 treatments to 2 years post last treatment
  Evaluate duration of local control
Evaluate Objective Response Rate (ORR) | After first 6 weeks of treatment
  Evaluate the proportion of patients who have a partial or complete response to therapy.
Evaluate Progression Free Survival | Post first 6 treatments to 2 years post last treatment
  Evaluate the length of time during and after the treatment that the subject lives with the disease but it does not get worse.
Evaluate Overall Survival | Post first 6 treatments to 2 years post last treatment
  Evaluate the length of time subjects stay alive from the date of first treatment.
PK Profile (C max) of Methoxsalen | First 6 weeks of study
  Establish C max of methoxsalen when given as an intra-tumoral injection
PK Profile (AUC) of Methoxsalen | First 6 weeks of study
  Establish AUC of methoxsalen when given as an intra-tumoral injection

CONTACTS AND LOCATIONS:
Overall Officials: William Eward, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Sibley Hospital - Johns Hopkins University, Washington D.C., District of Columbia
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Prisma Health, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported after deidentification for researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after the article publication to 36 months following article publication
Access Criteria: Proposals should be directed to smclaughlin@immunolight.com or lwood@immunolight.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 36 months on a third party website.